CLINICAL TRIAL: NCT03477786
Title: Blood Pressure Control to Reduce Renal Risk for Type 2 Diabetes Mellitus
Brief Title: Blood Pressure Control for Type 2 Diabetes
Acronym: BM4DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PH-107-PP-21
Record Dates: First submitted 2018-03-11; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tight BP (Active Comparator): Interventions: anti-hypertension drug prescription by physician and case management by health educator.
  Blood pressure is targeted at 120/80 mmHg in the tight BP control group.
  Interventions: Combination Product: drug adjustment and behavioral modification
- usual BP (Placebo Comparator): Interventions: The physicians follow their usual care patterns to prescribe anti-HT drugs.
  Blood pressure is targeted at < 140/90 mmHg in the usual BP control group.
  Interventions: Combination Product: drug adjustment and behavioral modification

INTERVENTIONS:
Combination Product: drug adjustment and behavioral modification — anti-hypertension drug prescription by physician and case management by health educator

SUMMARY:
The BP4DM study was initiated as a prospective randomized controlled trial to investigate the renal protection effect for tight blood pressure control for Taiwanese T2DM patients without previously diagnosed CV events. We set our primary outcome for the prevention of microalbuminuria development. The secondary outcomes include mortality, annual renal function declining rate, and development of cardiovascular events. The recruitment period for the RCT trial is from 2013 Oct to 2019 Dec. In addition, we also intend to continuously follow up all our recruited hypertensive diabetes patients for at least 10 years to observe their clinical outcomes including cardiovascular, renal, retinal outcomes and mortality.

DETAILED DESCRIPTION:
The evidence from previous literature shows importance of the blood pressure control in T2DM. About 20% (16-29%) reduction in microalbuminuria development can be reached by continuously lowering blood pressure level from 154/87 mmHg to 144/82 mmHg (the UKPDS), to 134.7/74.8 mmHg (the ADVANCE study), and even to 119.3/64.4 mmHg (the ACCORD study). However, several limitations are also inherent in the above well-known studies. First, most of the recruited participants previous trials were Caucasians. Although 3293 Chinese patients were recruited in the ADVANCE study, they only accounted for 29.6% of total enrollees in that trial. The representative of Asian population is inadequate. There is also lack of domestic evidence-based guideline designated for Taiwanese T2DM patients in optimizing their blood pressure control. In addition, some characteristics in Asian T2DM population are different from what have been observed in the Caucasian T2DM patients. For example, there is BMI discrepancy between T2DM in Western and Eastern countries, more ACEi/ARB side effects (e.g., cough) observed in Asian population, and the possible difference in CKD/ESRD incidence in T2DM between different ethnic groups.

Moreover, the enrollees in most well-known trials (e.g., ADVANCE and ACCORD studies) were those who suffered from at least one cardiovascular risk factor for secondary prevention. To our best knowledge, there is no study designed to evaluate effectiveness of blood pressure control for T2DM patients without previous CV events. Therefore, we initiated a prospective randomized controlled trial to investigate the renal protection effect for tight blood pressure control for Taiwanese T2DM patients without previously diagnosed CV events. We set our primary outcome for the prevention of microalbuminuria development to partly respond to the urgent need for this society in solving the huge burden caused by the high incidence and prevalence of diabetic nephropathy in Taiwan.

The study includes two parts: (1) a RCT trial, (2) an observational cohort study. The recruitment period of this study is from 2013 Oct to 2019 Dec. The RCT trial will be ended in 2019 Dec. In addition, we also intend to continuously follow up all our recruited hypertensive diabetes patients for at least 10 years to observe their clinical outcomes including cardiovascular, renal, retinal outcomes and mortality (the part of the observational cohort study).

ELIGIBILITY:
Inclusion Criteria (for both RCT trial and observational cohort study):

* type 2 DM with hypertension

Exclusion Criteria (for both RCT trial and observational cohort study):

* ACR>300 mg/g
* prior history of severe CV events (e.g., MI, stroke, heart failure>NYHA functional class III)
* dialysis, blindness, amputation, liver cirrhosis, cancer under active treatment
* pregnant women
* proteinuria which is unrelated with diabetes
* urinary tract stone > 0.5 cm

Stricter Exclusion Criteria (for RCT trial only):

* unstable BP (SBP>160 or DBP>100)
* unstable glycemic control (HbA1c>10%)
* K>5.0 meq/L

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-10-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
development of microalbuminuria | up to 10 years
  indicator of microalbuminuria: urine ACR

SECONDARY OUTCOMES:
mortality | up to 10 years
  all-cause mortality and CV-specific mortality
annual renal function declining rate | up to 10 years
  indicator of renal function: eGFR assessed by CKD-EPI formula
development of cardiovascular events | up to 10 years
  cardiovascular events include MI, heart failure, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Cheng Hsu, DrPH, Principal Investigator — National Health Research Institutes, Taiwan
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Min-Sheng General Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the trial is completed
Access Criteria: contact the principal investigator for data application